CLINICAL TRIAL: NCT03689569
Title: Effects of Prebiotic Supplementation and Exercise on Inflammatory Markers, Vascular Function, Cognition, and Mental Well-being in Pre-Dialysis Kidney Patients
Brief Title: Effects of Prebiotic Supplementation and Exercise on Inflammatory Markers, Vascular Function and Cognition in CKD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Springfield College (Other)
Responsible Party: Principal Investigator, Samuel A. Headley, Professor Exercise Science & Sport Studies, Springfield College
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Prebiotic study
Record Dates: First submitted 2018-09-19; First posted 2018-09-28 (Actual); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: Chronic Kidney Diseases
Keywords: microbiome; inflammation; resistant starch; exercise training
MeSH Terms: conditions — Renal Insufficiency, Chronic; Inflammation | interventions — Resistant Starch; Exercise; Starch

STUDY DESIGN:
Intervention Model Description: An Intention-To-Treat design will be used in this study. Effects of treatment on all dependent variables will be assessed by a 2 (prebiotic supplement or control) by 2 (aerobic exercise or control) by 3 (time) mixed factor ANOVA
Who Masked: Participant, Investigator
Masking Description: This will be a double blind study. Neither the participant nor the investigator will know what substance (resistant starch or corn starch) the participants will be consuming.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Exercise (Experimental): Exercise only: Patients randomized to this group will receive a placebo (corn starch) and be given 16 weeks of personal training.
  Interventions: Behavioral: Exercise
- Resistant Starch (Experimental): Resistant starch only: Patients randomized to this group will receive 30 g of resistant starch daily for 16 weeks. They will not be given an exercise training
  Interventions: Dietary Supplement: Resistant starch
- Exercise & Resistant Starch (Experimental): Exercise & resistant starch: Patients assigned to this group will do 16 weeks of personal training and they will be supplemented with 30 g of resistant starch daily for the 16 week period
  Interventions: Dietary Supplement: Resistant starch; Behavioral: Exercise
- Starch (Placebo Comparator): Corn starch only: Patients assigned to this group will not be given and exercise program and they will receive the placebo for 16 weeks
  Interventions: Behavioral: Starch

INTERVENTIONS:
Dietary Supplement: Resistant starch — Patients will receive 30 grams of resistant starch daily for 16 weeks or a placebo in a double blind fashion
  Arms: Exercise & Resistant Starch; Resistant Starch
Behavioral: Exercise — Patients randomized to the exercise group will train aerobically for 16 weeks at a moderate exercise intensity
  Arms: Exercise; Exercise & Resistant Starch
Behavioral: Starch — Patients will be given 30 grams of corn starch
  Arms: Starch

SUMMARY:
The study is primarily designed to examine the effect of 16 weeks of prebiotic supplementation (resistant starch)and moderate intensity aerobic training on markers of inflammation in stage 3-4 patients with chronic kidney disease.

DETAILED DESCRIPTION:
The primary aim of the proposed study is to determine whether the consumption of a prebiotic supplement (resistant starch) coupled with moderate intensity endurance training over 16 weeks leads to reductions in key inflammatory markers in stage 3-4 predialysis CKD patients and whether this reduction is associated with favorable changes in vascular function and indicators of stress and emotional reactivity.

The investigators hypothesize that supplementation with the prebiotic (resistant starch) will lead to normalization of the microbiome of our sample of patients with chronic kidney disease (CKD) and reduce key markers of inflammation. Reductions in these biomarkers will be associated with favorable changes in cardiovascular variables along with indices of stress and emotional reactivity. Moderate intensity aerobic training will have an additive anti-inflammatory effect along with the consumption of the resistant starch.

ELIGIBILITY:
Inclusion Criteria:

* stage 3-4 of CKD (GFR 15-59 ml/min/1.73m2),
* ages of 30-75 years old,
* Must be capable of complying with and following the study protocol(diet and exercise)
* Must be capable of independently giving informed consent

Exclusion Criteria:

* kidney transplant
* currently in a structured exercise program
* on antibiotic therapy within the last month
* On a probiotic or prebiotic supplement within the last month
* a GI disorder that prohibits the use of resistant starch (ie. high-amylose corn starch, which resists digestion
* HIV positive
* gastric by-pass surgery
* clostridium difficile
* marijuana user
* lupus
* rheumatoid arthritis
* Hepatitis C
* Post-traumatic stress disorder
* deep vein thrombosis
* pancreatitis

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-09-18 (Actual); Primary Completion 2021-05-31 (Estimated); Study Completion 2021-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in hs CRP | baseline and after 16 weeks
  hsCRP
Change in TNF alpha | Baseline and at week 16
  TNFalpha
Change in IL6 | Baseline and at week 16
  IL6
Change in IL10 | Baseline and at week 16
  IL10
Change in MCP1 | Baseline and at week 16
  MCP1

SECONDARY OUTCOMES:
Change in vascular function | Baseline, week 8 and week 16
  Pulse wave velocity
Change in microbiome composition | Baseline and after 16 weeks
  The composition of the microbiome will be assessed at baseline and after 16 weeks
Change in blood pressure | Baseline & after 16 weeks
  central blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Samuel A Headley, PhD, Principal Investigator — Springfield College
Locations (1):
- Springfield College, Springfield, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cooper TE, Khalid R, Chan S, Craig JC, Hawley CM, Howell M, Johnson DW, Jaure A, Teixeira-Pinto A, Wong G. Synbiotics, prebiotics and probiotics for people with chronic kidney disease. Cochrane Database Syst Rev. 2023 Oct 23;10(10):CD013631. doi: 10.1002/14651858.CD013631.pub2. PMID 37870148
- [Derived] Headley SA, Chapman DJ, Germain MJ, Evans EE, Hutchinson J, Madsen KL, Ikizler TA, Miele EM, Kirton K, O'Neill E, Cornelius A, Martin B, Nindl B, Vaziri ND. The effects of 16-weeks of prebiotic supplementation and aerobic exercise training on inflammatory markers, oxidative stress, uremic toxins, and the microbiota in pre-dialysis kidney patients: a randomized controlled trial-protocol paper. BMC Nephrol. 2020 Nov 26;21(1):517. doi: 10.1186/s12882-020-02177-x. PMID 33243160